CLINICAL TRIAL: NCT05087524
Title: Feasibility and Specificity of BinaxNOW for Diagnosis and Surveillance of Infection With SARS-CoV-2 in Schoolchildren
Brief Title: BinaxNOW for Evaluating Children for Infection With SARS-CoV-2 (COVID-19)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: changes in in-person schooling per COVID-19 pandemic
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-1521; Protocol Version 3/4/2021 (Other: UW Madison); A536756 (Other: UW Madison); philanthropic award (Other: American Family Children's Hospital)
Record Dates: First submitted 2021-10-18; First posted 2021-10-21 (Actual); Results first posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: SARS-CoV2 Infection; COVID-19
Keywords: diagnostic; diagnosis; schools; BinaxNOW; surveillance
MeSH Terms: conditions — COVID-19; Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- BinaxNOW Surveillance (Experimental): Participants will agree to the performance of nasal swabs samples to be used for diagnosis or screening. Samples will be obtained by research staff in the school setting. Madison Metropolitan School District (MMSD) has obtained a Clinical Laboratory Improvement Amendments (CLIA) waiver for collection of samples. When there is a positive test, a saliva sample will be collected for testing with a standard polymerase chain reaction (PCR) method. The standard PCR samples will be processed at University of Wisconsin (UW) Clinical Laboratory.
  Interventions: Diagnostic Test: BinaxNOW Ag Card

INTERVENTIONS:
Diagnostic Test: BinaxNOW Ag Card — A nasal swab specimen is collected from the participant, 6 drops of extraction reagent from a dropper bottle are added to the top hole of the swab well. The participant sample is inserted into the test card through the bottom hole of the swab well, and firmly pushed upwards until the swab tip is visible through the top hole. The swab is rotated 3 times clockwise and the card is closed, bringing the extracted sample into contact with the test strip. Test results are interpreted visually at 15 minutes based on the presence or absence of visually detectable pink/purple colored lines.

SUMMARY:
This is a study of the BinaxNOW Covid-19 Ag Card as a method to rapidly identify SARS-CoV-2 infection in asymptomatic children, teachers, and other school staff for exclusion. 240 students and 80 teachers in the Madison Metropolitan School District (MMSD) will be enrolled and can expect to be on study for up to 8 weeks.

DETAILED DESCRIPTION:
The overall purpose and research goal of this project is to understand how the virus SARS-CoV-2 is spread in the K-8 setting, decrease secondary cases of COVID-19, improve attendance and educational opportunities for children, teachers and other school staff, and decrease time away from work for parents (with threat of loss of employment and other benefits).

The investigators hypothesize that prompt diagnostic testing for SARS-CoV-2 in symptomatic children and twice weekly surveillance of asymptomatic children (with appropriate exclusion of children with positive tests) will be effective as a strategy to achieve maximum attendance in school and minimal disruption of the associated workforce.

STEP 1: Determine feasibility of using BinaxNOW COVID-19 cards for surveillance of infection with SARS-CoV-2 in teachers, other school staff, and school children.

The specific aims are to determine:

* if it is feasible to obtain nasal samples to be used with the BinaxNOW COVID-19 for diagnosis of COVID-19 in children or teachers/other school staff.
* if it is feasible to obtain nasal samples twice weekly to be used with BinaxNOW COVID-19 for surveillance of infection with SARS-CoV-2.
* The specificity of positive tests for SARS-CoV-2 obtained for diagnosis or surveillance compared to traditional PCR diagnostic testing.

STEP 2: Determine effectiveness of prompt diagnostic testing and twice weekly surveillance for SARS-CoV-2 among children and school faculty/staff to reduce the rate of positive cases (symptomatic) of COVID-19 in an elementary school setting resulting in an ultimate decrease in absenteeism for students and an increase in attendance for their parents at the workplace.

This is a record of the pilot study (STEP 1).

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5 - 15 years inclusive
* Currently attending school K-8 at one of the designated schools of the Madison Metropolitan School District
* Teachers and other school staff aged 20-65 years

Exclusion Criteria:

* Children < 5 years or > 16 years
* Teachers and other school staff < 20 years or > 65 years

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-01-09 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen R Wald, MD, Principal Investigator — UW School of Medicine and Public Health
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Madison Metropolitan School District (MMSD) Student and Staff Participants were enrolled from January to April 2021.
Groups:
- BinaxNOW Surveillance: Participants will agree to the performance of nasal swabs samples to be used for diagnosis or screening. Samples will be obtained by research staff in the school setting. MMSD has obtained a Clinical Laboratory Improvement Amendments (CLIA) waiver for collection of samples. When there is a positive test, a saliva sample will be collected for testing with a standard polymerase chain reaction (PCR) method. The standard PCR samples will be processed at University of Wisconsin (UW) Clinical Laboratory.
  BinaxNOW Ag Card: A nasal swab specimen is collected from the participant, 6 drops of extraction reagent from a dropper bottle are added to the top hole of the swab well. The participant sample is inserted into the test card through the bottom hole of the swab well, and firmly pushed upwards until the swab tip is visible through the top hole. The swab is rotated 3 times clockwise and the card is closed, bringing the extracted sample into contact with the test strip. Test results are interpreted visually at 15 minutes based on the presence or absence of visually detectable pink/purple colored lines.
Period: Overall Study
Arm/Group | BinaxNOW Surveillance
Started | 65
Completed | 65
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- BinaxNOW Surveillance: Participants will agree to the performance of nasal swabs samples to be used for diagnosis or screening. Samples will be obtained by research staff in the school setting.
Arm/Group | BinaxNOW Surveillance
Number analyzed (Participants) | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22
  Between 18 and 65 years | 43
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Gender of participants not collected.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 65

OUTCOME MEASURES:

1. Primary Outcome: Number of Tests Taken Per Participant
Description: Feasibility BinaxNOW surveillance testing will be measured by the number of test taken per participant. Greater than 1 test per participant is an indicator of compliance with repeat surveillance testing.
Time Frame: up to 8 weeks
Measure: Mean (Standard Deviation); unit: tests taken
Arm/Group | BinaxNOW Surveillance
Number analyzed (Participants) | 65
tests taken | 5.11 (2.56)

2. Primary Outcome: Number of Positive SARS-CoV-2 BinaxNOW Tests Confirmed by PCR Testing
Description: The specificity of positive tests for SARS-CoV-2 obtained for diagnosis or surveillance compared to traditional PCR diagnostic testing.
Time Frame: up to 5 weeks
Measure: Number; unit: positive tests
Arm/Group | BinaxNOW Surveillance
Number analyzed (Participants) | 65
positive tests | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were not collected.
Description: Adverse events data collection was not part of this protocol.
Arm/Group | BinaxNOW Surveillance
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
This study was terminated early due to changes in in-person schooling per COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2021-03-04): https://cdn.clinicaltrials.gov/large-docs/24/NCT05087524/Prot_001.pdf